CLINICAL TRIAL: NCT06651918
Title: The Effect of Yoga Practice on Fatigue Quality of Life and Symptoms in Children With Cancer
Brief Title: Effects of Yoga on Children With Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Eda Kalayci, pediatrıc nurse, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: ErciyesEKalayci38
Record Dates: First submitted 2024-04-04; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Cancer
Keywords: children with cancer; yoga; fatique; quality of life; symptoms of cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga practise (Experimental): For the experimental study, the researcher will contact the participants to be included in the study and the intervention (yoga group) and control groups will be randomly created. The participants will be informed about the study by the researcher and their voluntary consent will be obtained. The researcher will provide information about the Identifying Characteristics Form for Children Diagnosed with Cancer and Their Families, the Quality of Life Scale for Children (PedsQL) and the Memorial Symptom Assessment Scale to be used in the study. The survey and scales will be applied to each participant individually one day before yoga. Then, the Yoga Group will be applied 3 sessions per week, 3 weeks in a row, each session will be 30 minutes. The researcher will repeat the survey and scale questions that he asked the participants before they started yoga at the end of the 3 weeks.
  Interventions: Behavioral: yoga practise
- survey group (No Intervention): No intervention will be made to the children in this group, only survey and scale questions will be applied.

INTERVENTIONS:
Behavioral: yoga practise — For the experimental study, the researcher will contact the participants to be included in the study and the intervention (yoga group) and control groups will be randomly created. The participants will be informed about the study by the researcher and their voluntary consent will be obtained. The researcher will provide information about the Identifying Characteristics Form for Children Diagnosed with Cancer and Their Families, the Quality of Life Scale for Children (PedsQL) and the Memorial Symptom Assessment Scale to be used in the study. The survey and scales will be applied to each participant individually one day before yoga. Then, the Yoga Group will be applied 3 sessions per week, 3 weeks in a row, each session will be 30 minutes. The researcher will repeat the survey and scale questions that he asked the participants before they started yoga at the end of the 3 weeks.
  Arms: yoga practise

SUMMARY:
This study was planned as a randomized controlled experimental study with a pre-test-post-test design to determine the effect of yoga practice accompanied by a specialist yoga instructor on fatigue, quality of life and symptom control in children diagnosed with cancer between the ages of 8-12.The main questions it aims to answer are:

1. Does yoga practice applied to children diagnosed with cancer reduce fatigue in children?
2. Does yoga practice applied to children diagnosed with cancer affect their quality of life?
3. Does yoga practice applied to children diagnosed with cancer affect the symptoms experienced by children?

Before and after yoga practice, children diagnosed with cancer will answer survey and scale questions about fatigue, quality of life and symptoms.

DETAILED DESCRIPTION:
Cancer is among the major health problems all over the world. Every year, 400 000 children are diagnosed with cancer all over the world and 3500 children are diagnosed with cancer every year in our country. It is estimated that the number of children diagnosed with cancer will increase exponentially every year. In addition to this increase in the incidence of childhood cancers, developments in medicine and technology in recent years have enabled the life expectancy of children diagnosed with cancer to extend. However, cancer and its treatment cause physiological and psychosocial problems that can negatively affect the lives of children diagnosed with cancer. Symptoms such as pain, fatigue, sleep problems, nausea/vomiting, loss of appetite, physical activity intolerance, stress/anxiety are common in children with cancer, depending on the disease and its treatment, and they negatively affect the quality of life of children In order to reduce the negative effects of symptoms caused by cancer and its treatment, it is important to separately evaluate and address the quality of life of children diagnosed with cancer and factors such as sleep, fatigue, stress and physical activity, which constitute the quality of life components. It is recommended to use complementary treatment methods, including mind-body practices, to improve the quality of life of children diagnosed with cancer and to reduce the symptoms and effects that may occur. Complementary treatment methods include massage, acupuncture, breathing exercises, relaxation techniques, laughter therapies and yoga. Children's yoga, which has been used in children with cancer in recent years, is defined as physical activity that provides strength, balance and movement in children, as well as activities that increase awareness through breathing work. It has been determined that yoga activity has positive effects on the physiological and psychological measurements and quality of life of children with cancer.

The fact that yoga activity can be done in any area without the need for any materials provides an advantage for children diagnosed with cancer. The play and activity needs of children with cancer who are isolated due to cancer and its treatment must be met under safe conditions. Children's yoga, performed with simple and fun movements in the hospital room, can increase the activity of the child with cancer and meet the need for play and activity. It may also help the child diagnosed with cancer to shift the focus away from the disease and the negative effects that the disease may have caused. Improving the quality of life of children diagnosed with cancer, reducing/controlling the symptoms caused by cancer or its treatment, and planning and implementing new coping methods are among the main goals of pediatric oncology nurses. Although there are studies on the effects of yoga practice on children with cancer in the literature review, there are limited studies on this subject in our country. In line with all these, this research was planned as a randomized controlled experimental study to determine the effect of yoga practice on the symptoms, fatigue and quality of life experienced by children diagnosed with cancer.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be between the ages of 8-12,
* He/she must not have a chronic or genetic disease other than cancer,
* He/she must not have a physical, mental or neurological disability,
* The participant must have a mother who is at least a primary school graduate,
* The participant must be able to speak and understand Turkish,
* Both the participant and his/her parents must be open to communication and cooperation,
* Participants will be included in the study if both the participant and his/her parents agree to participate in the study voluntarily and give verbal and written consent.

Exclusion Criteria:

- Participants who do not want to participate in the study or who want to leave the study, who have communication difficulties, and who have solid tumors (Osteosarcoma, Ewing sarcoma, etc.) that prevent them from doing yoga will be excluded from the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Inventory for Children (PedsQL) | At the beginning yoga and after three weeks ; survey and scale questions will be applied by the researcher. In addition, in the statistical analysis section of the research, correlation and regression analysis will be conducted between the measure
  The scale, developed by Varni and his colleagues in 2001 and adapted into Turkish by Çakın-Memik et al. (2007), questions the quality of life of children in the areas of physical, emotional, social and school functionality.
Memorial Symptom Assessment Scale (7-12 years old) | At the beginning yoga and after three weeks ; survey and scale questions will be applied by the researcher. In addition, in the statistical analysis section of the research, correlation and regression analysis will be conducted between the measure
  The scale, which was developed by Collins et al. in 2002 for use in children with oncology between the ages of 7 and 12, was adapted into Turkish by Şenol and Efe (2022).It is used to evaluate symptoms of pain, numbness, sadness, nausea, pruritus, anxiety, loss of appetite, and insomnia experienced by pediatric oncology patients in the past two days.
Fatigue Assessment Scale for Pediatric Oncology Patients Aged 7-12 | At the beginning yoga and after three weeks ; survey and scale questions will be applied by the researcher. In addition, in the statistical analysis section of the research, correlation and regression analysis will be conducted between the measure
  The Fatigue Assessment Scale for Pediatric Oncology Patients Aged 7-12, developed by Kudubeş, Bektaş and Uğur in 2019, consists of 27 items and 3 sub-dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Erdem, Prof., Study Director — TC Erciyes University

IPD SHARING:
Plan to Share IPD: No